CLINICAL TRIAL: NCT00180557
Title: Analyse Der Unterschiede Zwischen Aktiv-fixierenden Und Passiv-fixierenden Stimulations-Elektroden Hinsichtlich Implantationsdauer Und Elektrischer Parameter
Brief Title: Austria Study - Analysis of Difference Between Active and Passive Fixation Leads
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guidant Corporation (Industry)
Responsible Party: Rainer Habeler, Guidant Austria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Austria Study v. 1.2
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2007-12

CONDITIONS: Bradycardia; Heart Block; Sick Sinus Syndrome
MeSH Terms: conditions — Bradycardia; Heart Block; Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active fixation lead (Experimental): Active fixation lead was implanted
  Interventions: Device: Flextend II, Fineline 2, Fineline Atrial J, Selute Picotip
- Passive fixation lead (Active Comparator): Passive fixation lead was implanted
  Interventions: Device: Flextend II, Fineline 2, Fineline Atrial J, Selute Picotip

INTERVENTIONS:
Device: Flextend II, Fineline 2, Fineline Atrial J, Selute Picotip

SUMMARY:
In this study the difference between screw in leads actively fixed in the septum and tined leads passively fixed in the apex concerning electrical parameters and implantation time will be evaluated. In addition the influence of the stimulation location by type of lead on QRS width, ejection fraction and NYHA class will be evaluated using and electrocardiogram and echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

Age < 18 years, indication for pacemaker implantation according to current guidelines, written consent of the patient

Exclusion Criteria:

Live expectancy < 6 months, pregnancy or women without contraception in birth bearing age, inability or refusal to sign consent form, simultaneous participation in another clinical trial, contraindication for any procedure required during pacemaker implantation, patients who need other pacemaker systems including pacing leads than those required by the protocol, heart failure (LVEF <35%, QRS-Width>150ms), functional (rate dependent) bundle branch bloc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
QRS width
Ejection fraction
NYHA class

CONTACTS AND LOCATIONS:
Overall Officials: C Nimeth, MD, Principal Investigator — Krankenhaus der barmherzigen Schwestern Ried im Innkreis
Locations (1):
- Krankenhaus der barmherzigen Schwestern, Ried im Innkreis, Austria